





# **Huntington's Disease Young Adult Study 2.0**

7<sup>th</sup> September 2023





# **HD-YAS 2.0**

# Huntington's Disease Young Adult Study 2.0

Information Sheet and Informed Consent Form

# **Control Participant**

Version 2.1, 7<sup>th</sup> Sept 2023(IRAS number: 303499, EDGE (sponsor) number: 145646, REC ref: 22/LO/0058)

#### I. Part I

#### 1. Invitation Paragraph

You are being invited to participate in a research study named Huntington's Disease Young Adult Study 2.0 (HD-YAS 2.0). You have been invited to take part because you completed YAS 1.0 or because you have been identified as a new eligible participant. Before you decide whether to participate it is important for you to understand why the research is being done and what it will involve. Please take time to read the following information carefully and discuss it with others if you wish. Ask us if there is anything that is not clear or if you would like more information.

#### 2. What is Huntington's Disease?

Huntington's disease (HD) is an inherited neurodegenerative disease. A faulty gene causes the buildup of a toxic protein - mutant huntingtin - which damages brain cells, leading to problems with movement, thinking and behaviour. The faulty gene can be passed down within families, a person whose parent has HD is born with a 50-50 chance of inheriting the faulty gene. Anyone with a family history of HD can choose to have a predictive genetic test, which means they can find out whether they have the faulty gene or not, and therefore, whether they will go on to develop the disease or not.

# 3. What is the purpose of the study?

The HD-YAS 1.0 study revealed that, although function was completely normal, there was some evidence of subtle early changes in gene carriers decades from developing the disease. The purpose of HD-YAS 2.0 is to determine whether there is any change over time in these early disease signs. The 131 participants who took part in HD-YAS 1.0 are being invited back to undergo similar assessments so we can look at what has changed. New participants are also being included to account for participants from the first study who may not want to participate again. This will help us to guide the use of any potential future treatments, so that they can be given at the earliest and most effective time in order to prevent or treat HD disease progression.





# 4. Do I have to take part in this study?

No, your participation in this study is completely voluntary. You are free to choose whether or not to participate in this study. If you decide to participate, you can change your mind and withdraw from this study at any time, for whatever reason. You are not required to give any reason for your decision on whether or not to participate in this study or, if you decide to participate, for your decision to withdraw from this study. Deciding not to participate in this study, or deciding to withdraw from this study will not affect the current or future care that you would otherwise expect to receive.

# 5. What will happen to me if I take part in this study?

If you agree to take part, you will be asked to attend two study visits at the National Hospital for Neurology and Neurosurgery (NHNN) London, roughly 2 years apart, each of which will last a whole day or two/ three days if you choose to take part in the optional CSF and matching blood collection and the optional 7T MRI and MEG scans. The visit may involve an overnight stay, depending on how far you have to travel and there will be plenty of time for refreshments, lunch and breaks. After the visit, we ask you to complete some more questionnaires online either at home or after CSF collection. If you choose to take part in the CSF collection then a few days after the visit you will also receive a telephone follow-up to check how you are after this procedure. More information about what will happen on each study day can be found it Part 2 of this information sheet.

## 6. Who is organising HD-YAS?

This research is being organised by Professor Sarah Tabrizi (Principal Investigator), Professor of Clinical Neurology, Honorary Consultant Neurologist and Director of UCL Huntington's Disease Centre and is sponsored by University College London. The HD-YAS 2.0 study is funded by the Wellcome Trust. CSF collection is funded by CHDI Foundation Inc., a not-for-profit foundation that only works on HD.

#### II. PART 2

#### 1. How many participants will be involved?

Up to 161 participants will be included in this study – 131 who completed the original HD-YAS study (64 people who carry the HD gene, but do not show any signs of the disease and 67 control participants) and up to 50 new participants (25 people who carry the HD gene, but do not show any signs of the disease and 25 control participants). A control participant is a person who does not carry, and is not at risk of carrying the genetic mutation that causes HD.

## 2. Study Visits

The study consists of two study visits, which will take place two years apart. Each of these study visits will be exactly the same and be organised as follows:

#### Day 1 – Consent, MRI, Cognitive and Emotional Assessments

At the study visit, you will have a number of assessments, performed by experienced professionals.

HD Young Adult Study 2.0, EDGE (Sponsor) number: 145646, IRAS number: 303499, Control PIS/ICF, Version 2.1, 7th Sept 2023 







You are encouraged to eat a good breakfast before the session starts. Breaks will be included throughout the day but you may also request break sessions as needed. You can find more information about each procedure further on in this information sheet. You will need to be fluent in English to complete the cognitive assessments. Your height and weight will also be measured.

A schedule of the study visit and estimated times are shown below:

| Time | Assessment Type | Duration |
|---|---|---|
| 9:00 | Informed Consent for HD-YAS 2.0, including for CSF collection and optional imaging acquisition if applicable. | 30 min |
| 9:30 | Clinical review and blood sample | 45 min |
| 10:15 | Break | |
| 10:45 | Cognitive and Emotional Assessments | 115 min |
| 13:00 | LUNCH | |
| 14:00 | MRI scan | 90 min |
| 15:30 | BREAK | |
| 16:00 | HD core assessment battery | 60 min |
| 17:00 | END OF STUDY VISIT | |

Overnight hotel stay near study site following Day 1 assessments. Fasting from midnight for CSF and blood collection (water only)

# Day 2 - CSF collection

You will arrive at the site sometime between 8:00 and 9.00 am. You will need to be fasted from midnight the night before, drinking only water and the study doctor will make sure it safe to go ahead with the lumbar puncture. Following the sample collection you will be asked to lie flat for up to an hour. Breakfast will also be provided for you.

A schedule of the study visit and estimated times are shown below:

| 8:00 - 9:30 | Optional - CSF and blood collection | 45 min, plus resting time |
|---|---|---|
| 9:30 - 10:15 | Neuropsychiatric self-report assessments | 45 min |

HD Young Adult Study 2.0, EDGE (Sponsor) number: 145646, IRAS number: 303499, Control PIS/ICF, Version 2.1, 7th Sept 2023 







1-3 days after CSF collection

Telephone follow-up to check for adverse events following the optional CSF collection. Follow-up details to be entered on to a paper record by researcher.

#### Additional 7T and MEG collection

You will arrive at the The Wellcome Centre for Human Neuroimaging and a radiologist will ask you some questions to make sure it is safe to scan you. The MEG task will then be explained to you and you will have a chance to practice the task outside the scanner before you undergo the scan. After a break you will then undergo the 7T MRI scan.

A schedule of the study visit and example times are shown below:

| Time | Assessment Type | Duration |
|-------|-------------------|-----------|
| 13:00 | Safety screening | 30mins |
| 13:30 | MEG Task practice | 30mins |
| 14:00 | MEG Scanning | 60-90mins |
| 15:00 | BREAK | |
| 15:30 | 7T MRI | 60 mins |

#### 3. Procedures

## **Blood Sample Collections**

We will collect up to 60 mls of blood (approximately 12 tablespoons) from a vein in your arm in the usual way. The skin around the injection site will be cleaned and a small needle will be inserted to draw blood. This procedure is quick, typically taking just a few minutes to do and will be performed by an experienced and trained member of the research team.

- Your blood will be used to look for biomarkers a biomarker is something we can measure that helps us to better understand a disease. We intend to relate any changes we may see in biomarkers to any early changes we may see in the brain and functioning. As a control participant it is valuable to obtain these samples so we can compare the results to those obtained from HD gene carriers to help understand the significance of any results. This information does not reveal anything of clinical significance to you. The result of the tests will not be made available to you.
- > If you are participating in the CSF collection we will also use your blood to check safety markers to make sure it is safe to collect CSF from you.

There is a small risk of discomfort, bruising or bleeding associated with having a blood sample taken. Sometimes people can feel faint or light-headed during or shortly following blood collection. You will

HD Young Adult Study 2.0, EDGE (Sponsor) number: 145646, IRAS number: 303499, Control PIS/ICF, Version 2.1, 7th Sept 2023 





# University College London Hospitals **NHS**



be given plenty of time to rest if you feel unwell, until you feel better. There is also a small risk that a clot may form at the site of needle puncture and infections may occur, but these are rare.

### **Cognitive and Emotional Tasks**

You will spend about two hours doing some thinking tasks, which will include for example, trying to remember the location of shapes on the screen or find a pattern in a sequence. As well as emotion tasks like detecting emotions on faces in pictures or rating your feelings in response to a set of moral scenarios. There will be a number of different tasks to assess different areas of thinking and emotion. The tasks are performed using a computer but you do not need to have any knowledge of computers in order to do them. You should bring reading glasses if you require them.

#### 3T MRI scan

MRI is a painless and safe technique that can provide detailed pictures of the brain. It uses a magnetic field and radio waves, together with an advanced computer system to build up a 3D image.

The MRI scanner is like a tunnel about 1.5 metres long, surrounded by a large circular magnet. You lie on a couch which then slides into the scanner. The scanner will produce loud noises; this is normal and should not worry you. However, you will be provided with earplugs and/or headphones. During the MRI, the operator will be able to speak to you, hear you, and observe you at all times through a window and a 2-way microphone communication system.

MRI does not use any harmful radiation, it is painless and there are no known side-effects or cumulative risks. However, the powerful magnetic field of the MRI scanner can attract certain metallic objects, causing them to move suddenly and with great force towards the centre of the MRI machine. This may pose a risk to anyone in the way of the object. Therefore, great care is taken to prevent such objects e.g. watches, jewellery, hair pins and items of clothing that have metallic threads or fasteners from entering the MRI room. The MRI facility safety assessment requires MRI staff and radiologist to ask about the presence of metallic implants and tattoos etc. Research suggests that heating and pulling can occur with older tattoos, which may contain small quantities of metal. Therefore, participants with tattoos are sometimes excluded from MRI scans unless special precautions are taken.

Female participants: If you are pregnant or think that you could be pregnant, you must notify the MRI operator or radiologist during the safety assessment. Depending on the outcome of the safety assessment, you may not be able to have the scan.

The scan lasts up to 90 minutes but takes place in several parts, up to 15 minutes each. You will need to keep still during each part of the scan but can move a little between parts.

#### **HD Core Assesment Battery**

During your study visit we will ask questions about your medical history, your current health and any medications you are taking. We will measure your height and weight. We also will conduct tests to see how well you move, think, remember things, perform daily tasks, and behave – all behaviours which may be affected by HD. The examination should take about 60-75 minutes.

## **Patient Reported Neuropsychiatric Questionnaires**

You will be asked to complete 10 self administered, short questionnaires either after the CSF collection or at home between 1 and 7 days after the study visit. These questionares will take approximately 4

HD Young Adult Study 2.0, EDGE (Sponsor) number: 145646, IRAS number: 303499, Control PIS/ICF, Version 2.1, 7th Sept 2023 





# University College London Hospitals **NHS**



minutes each to complete and they will gather information about a a collection of symptoms including sleep, mood, motivation, anxiety and depression. These are common symptoms that can occur in anyone in the population at any time. We will ask you to complete these questionnaires online either at home or after CSF collection. You will be provided with information on how to answer these questionnaires and return them to us.

# **HD-YAS 2.0 Optional Component - CSF and Blood Collection**

In addition to the main part of this study, as described above, there is an optional part where we will collect cerebrospinal fluid (CSF), the fluid surrounding the brain and spinal cord. This provides information about the brain and the nervous system that is impossible to obtain in any other way.

An optional blood sample will also be collected to match the CSF collection.

# What Will Happen to Me if I Take Part?

We will ask you to donate up to 20ml of CSF (approximately 4 teaspoons) by lumbar puncture. Once the CSF collection has been completed, approximately 50 ml of blood (the same volume as 10 teaspoons) will be taken from a vein in your arm.

#### Do I Have to Take Part?

You can choose whether or not you want to take part in the CSF collection, it is entirely optional and you can choose to take part in one, all or no aspects of the study. If you choose to participate in the optional CSF collection you will be asked to provide specific consent.

#### **Proceedures and Study Visits**

You will be invited to attend a second study day as outlined in Section 2- Study Visits. Overnight accomadation will be arranged for you in a nearby hotel if needed.

#### **Lumbar Puncture**

A lumbar puncture is a medical procedure where a very thin needle is inserted into the lower back to collect CSF fluid. It is a very common procedure that typically takes around 30 minutes to perform.

At the start of the procedure you will be asked to lie on your side with your knees pulled up and your chin tucked downward. A pillow will be placed between your knees. The skin around your lower back area is cleaned and local anaesthetic will be injected, this stings for a couple of minutes, then the skin goes numb. After a couple of minutes a very thin needle will be inserted into your lower back to collect the CSF, occasionally it may be necessary to try again in a different spot, or for you to sit upright, to find the right place and collect the fluid. Although the local anaesthetic makes the skin go numb some people can still experience some pain during the procedure. You are free to ask for the procedure to be stopped at any time.

Following the sample collection you will be asked to lie flat for up to an hour. The entire procedure of collecting CSF and blood should take about 20-45 minutes, not including the resting period. The study site staff will check to see how you are doing during the resting period. When you are ready to leave, you will be given instructions on follow-up care.

HD Young Adult Study 2.0, EDGE (Sponsor) number: 145646, IRAS number: 303499, Control PIS/ICF, Version 2.1, 7th Sept 2023 







#### **Blood Collection**

Once the CSF collection has been completed, approximately 50 ml of blood (the same volume as 10 teaspoons) will be taken from a vein in your arm in the same manner as describe above.

## Follow-Up Call: 1 to 3 Days after optional CSF Collection

We will call you 1 to 3 days after the CSF and Blood collection to ask you how you are feeling and if you have experienced any medical conditions or symptoms since your visit.

#### What discomforts and risks are involved?

# Some of the possible **discomforts of CSF collection** include:

- The anaesthetic will sting when first injected.
- You may feel a pressure sensation when the needle is inserted.
- Some people experience brief pain, either in the back or down one leg, when the needle is close to the spinal fluid. This pain usually stops after a few seconds.
- You may experience some back pain following the CSF collection.
- You may experience a headache following the CSF collection. You will be given instructions on how to manage this if it occurs. The risk of headache is about 19%. Occasionally the headache doesn't go away on its own and a second hospital procedure called a "blood patch" may be recommended to help it resolve. This is rare - the chance is less than 1% overall.

#### Possible risks of CSF collection include:

- Hypersensitivity (allergic) reaction to the anaesthetic.
- Infection caused by the needle going through the skin. This is very rare; the risk is much less than
- Damage to the nerves in the lower back, which could cause numbness, pain or altered function in the legs, bowels, bladder or genitals. This may be caused directly by the needle or by blood leaking into the fluid. It is very rare (much less than 1 in 1,000).

# HD-YAS 2.0 Additional Component in Subset of Participants – MEG and 7T MRI

## Why have I been invited to undertake additional brain scans?

In addition to the procedure described above, there is another part of the study that a subset of participants will be invited to complete. We will invite 20 gene-carriers and 20 control participants. We will obtain images of the brain using Magnetoencephalography (MEG) imaging and 7 Tesla (7T) MRI. This produces more detailed, higher quality images which can detect more subtle changes.

You have been invited to take part in this additional component as you are known to tolerate MRI scanning well and you have donated CSF in the original YAS study.

## What Will Happen to Me if I Take Part?

We will ask you to attend another study day to undergo a MEG scan and a 7T MRI scan. You will also be shown how to play a computer game task that we will use during the MEG scanning.

### Do I Have to Take Part?

HD Young Adult Study 2.0, EDGE (Sponsor) number: 145646, IRAS number: 303499, Control PIS/ICF, Version 2.1, 7th Sept 2023 







# University College London Hospitals **NHS**



You can choose whether or not you want to take part in the MEG and 7T MRI, it is entirely optional and you can choose not to take part in it even if you are invited by the study team.

# **Procedures and Study Visits**

You will be invited to attend a third study day as outlined in Section 2- Study Visits. Overnight accommodation will be arranged for you in a nearby hotel if needed.

# Magnetoencephalography (MEG) scan

MEG is a painless and safe technique that measures magnetic fields produced by brain cell activity. It involves sitting in a specially constructed room while a helmet containing sensors is placed around your head. MEG does not use any harmful radiation and there are no known side effects or cumulative risks.

### **High-resolution 7T MRI scan**

High-resolution 7T MRI scanning is the same as the 3T MRI described above, except it uses stronger magnets, which allow us to obtain more detailed images of the brain. Some people scanned in MRI scanners, especially 7 Tesla scanners, may experience a mild dizzy sensation as they are moved into and out of the scanner. This is normal and the sensation starts to go away as soon as you are in the scanner. In order to minimise and avoid these effects, movement into the scanner is done slowly by an advanced MRI operator.

# 4. What must I keep in mind during this study?

During the time of this study, you are being asked to follow all instructions that the study physician and study team give you. If you choose to partake in the CSF and blood collection you should also follow instructions regarding follow-up care after the CSF and blood collection which will be explained to you by the study doctor.

On the day of CSF and blood sampling visit you will be asked to not eat anything from midnight the night before until the CSF and blood collection has been completed.

If you are not feeling well or if you have had medications since your referral to us for the study or the telephone call to arrange your study visit you should inform the study team as soon as possible.

# 5. How will my samples and information be stored?

All the information we collect during the course of the research will be kept confidential and there are strict laws which safeguard your privacy at every stage.





We will need to use personal information from you and from your medical records for this project. This information will include your name, date of birth, contact details, MRI screening forms and, where applicable, GP letters, surgical notes and genotyping reports,. People will use this information to do the research or to check your records to make sure that the research is being done properly.

The personal information collected about you during this study will be entered via secure internet connections into a confidential database, called the Data Safe Haven, that is located on a secure server through the study sponsor, University College London. In addition, any paper copies of the data will be held securely in a locked cabinet, in a security-controlled office at the UCL HD centre. Access will be restricted to authorised personnel. The biological samples collected during this study will be stored in a repository at UCL Institute of Neurology for which Prof Tabrizi is the custodian.

We will not put your name, address or any other information that could directly identify you on the information and biological samples you allow us to collect from you. Instead this will be coded with a subject ID or a Huntington's disease identifier (HDID), the unique 9 digit number created for you as part of your participation in the original HD-YAS study, or we will create this for you. The HDID is used to protect your identity and connect your clinical information and biological samples to other HD studies in which you may participate. Only the study site staff will be aware of your identity and be able to link the information and biological samples collected from you during this study. All information and biological samples collected will be stored in secure databases and repositories.

# 6. How will my samples and information be used and shared?

The coded information and/or coded biological samples collected from you may be used by Prof Tabrizi, her research team members, her appointed service providers, and her appointed partners from academic, not-for-profit and/or commercial research organisations, for the following purposes:

- To generate a CSF sample collection and a blood products sample collection for identifying and evaluating biomarkers and pathways that will enable the development of new treatments for HD.
- To check the quality of the information and biological samples collected from you during this study.
- To see how different possible medicines influence biological and chemical processes that might be important in HD or other diseases.
- To design and guide future research studies and clinical trials.
- To support and enable scientific discussion and research as follows: (1) to better understand HD or other diseases being studied, (2) that furthers the development of treatments for HD or other diseases or (3) that furthers biomedical research.

This may include the development of commercial products from which you will not benefit financially.

Your coded information and a portion of your coded biological samples will be shared with CHDI Foundation Inc. (CHDI), a not-for-profit foundation that only works on HD. CHDI will store your coded biological samples in a biological samples repository (storage facility) and your coded information in one or more electronic databases. CHDI may also share your coded information and coded biological samples with other researchers and service providers for the purposes already stated above.





To meet regulations or for reasons related to this study, Prof Tabrizi may also share this consent form and records that identify you and biological samples collected from you during this study with the following third parties:

- Representatives of organisations providing services in connection with this study, the organisation contracted to collect, maintain, and manage the information collected in this study alongside UCL; service providers engaged to check the accuracy of the information collected; and such other service providers as may be designated from time to time.
- Representatives of governmental and regulatory agencies

Prof Tabrizi, the study sponsor (UCL), CHDI and each of the organisations, researchers and services providers referred to above, may publish the results of their research, including coded information, in medical journals or present such results at meetings. However, your name, address or any other information that could directly identify will not be published.

The information and biological samples collected from you during this study will be used only for research purposes and will not be sold.

You can change your mind at any time about the storage and use of the biological samples collected from you during this study. Just contact Prof Tabrizi or a member of her research team, and let him or her know that you no longer want the biological samples collected from you during this study stored and such biological samples will be removed from the storage facility and destroyed. If any biological samples collected from you during this study have already been distributed for use, it may not be possible for us to locate and destroy them.

Any of the uses and activities described above may involve sending coded information and coded biological samples to other countries that may not have the same or as strict privacy laws as this country. However, given that only coded information or coded biological samples are sent, the risk of unintended disclosure of identifying information is low.

Whilst we do not want to cause alarm, we are required by the body governing Research Ethics Committee to let participants know what will happen to their samples and/or data if they were to lose capacity during the course of the study (or thereafter). Should you lose the capacity to consent during your participation, you will be withdrawn from the study by the research team, and we would like to ask your permission in advance to retain any CSF and/or blood samples collected prior to your withdrawal for use in HD research.

If you would like any further information about how we use your data, you can find out more:

- at www.hra.nhs.uk/information-about-patients/
- our leaflet available from www.hra.nhs.uk/patientdataandresearch
- by asking one of the research team
- by sending an email to the study manager on k.fayer@ucl.ac.uk, or
- by ringing us on 02031087483.
- 7. What other discomforts and risks are involved?





Any adverse medical events arising from your participation in this study will be followed up and treated as necessary by the study team.

### Assessments and questionnaires

When completing the clinical, behavioural and cognitive assessments for HD-YAS, you may experience low mood or psychological discomfort (such as stress or anxiety). If at any time you feel you could benefit from treatment or support, you may request to be referred for appropriate care. In the course of doing these questionnaires or tests you may also feel tired and/or irritable. If this happens please tell your doctor or a member of the research staff and ask them to allow you time to rest or stop the testing all together.

# Collection of private / personal information

We take great care to protect your personal information and all procedures are in compliance with the Data Protection Act 2018 and the General Data Protection Regulation (GDPR). However, there is a slight risk of accidental disclosure of information, or breach of computer security.

For more information you can read UCL privacy notice for Participants and Researchers in Health and Care Research Studies here: <a href="https://www.ucl.ac.uk/legal-services/privacy/ucl-general-privacy-notice-participants-and-researchers-health-and-care-research-studies">https://www.ucl.ac.uk/legal-services/privacy/ucl-general-privacy-notice-participants-and-researchers-health-and-care-research-studies</a>

UCL also has a data protection policy that sets out our commitment to the safeguarding of personal data processed by its staff and students and our stances on compliance with data protection legislation. This can be read here: <a href="https://www.ucl.ac.uk/information-security/sites/information-security/files/data-protection">https://www.ucl.ac.uk/information-security/sites/information-security/files/data-protection</a>

# **Unexpected findings**

We do not expect to find anything of medical significance for individual research participants as part of this study. The results of the tests will not routinely be conveyed to you. However, occasionally, an MRI scan, blood tests or a lumbar puncture can reveal an unexpected finding of possible medical importance. If this happens, we will let you know and, with your permission, inform your GP who will be able to take any necessary action through the usual NHS care pathways.

# 8. What are the benefits of taking part in HD-YAS?

You will not have any direct benefits from participating in this study. The results of this study may contribute to new knowledge of HD.

## 9. What are the alternatives to taking part?

You do not have to participate in this study. Choosing not to participate will not affect your current or future medical care at the National Hospital for Neurology and Neurosurgery.

## 10. Is there any payment or cost?

Your expenses, including meals and hotel (if applicable) incurred within the scope of your participation in this study will be covered. You will need to provide receipts for your expenses. We can usually help book travel and accommodation so you don't have to pay upfront. Please consult

HD Young Adult Study 2.0, EDGE (Sponsor) number: 145646, IRAS number: 303499, Control PIS/ICF, Version 2.1, 7<sup>th</sup> Sept 2023 





the study team before spending your own money, to make sure the expense will be refunded, as some items like train fares and hotel accommodation have limits on how much can be reimbursed.

In addition, participants that undergo the Lumbar Puncture for CSF sampling will receive compensation in the amount of GBP 200 after each sampling visit. This is to compensate you for the additional time and discomforts arising from CSF sampling.

# 11. What happens if I am injured or something goes wrong?

If you wish to complain, or have any concerns about the way you have been approached or treated as part of this study, you should contact Prof Tabrizi or a member of her team, who will do their best to address your concerns. The National Health Service or UCL complaints mechanisms are available to you. Please ask Prof Tabrizi or a member of her team if you would like more information on this.

UCL Hospitals Foundation Trust will provide medical care for any emergency medical problem that you may experience as a direct result of your participation in this research. You will not have to pay for this emergency care.

We will notify your GP that you are taking part in this study, unless you have told us that you would prefer that your GP is not made aware of your participation.

If you have health insurance, it is up to you to find out whether participation in this study may affect your insurance cover.

In the unlikely event that you are harmed by taking part in this study, compensation may be available. University College London (UCL) holds insurance against claims from participants for harm caused by their participation in this clinical study. Participants may be able to claim compensation if they can prove that UCL has been negligent. However, if this clinical study is being carried out in a hospital, the hospital continues to have a duty of care to the participant of the clinical study. University College London does not accept liability for any breach in the hospital's duty of care, or any negligence on the part of hospital employees. This applies whether the hospital is an NHS Trust or otherwise.

If you have concerns about any aspect of this study, you should call 020 3108 7480 and ask to speak to the researchers who will do their best to answer your questions.

If you remain unhappy and wish to complain formally, you can do this by contacting the Patient Advice and Liaison Service on 020 3448 3237 or write to UCLH Patient Advice and Liaison Service at the following address; PALS, Box 25, National Hospital for Neurology and Neurosurgery, Queen Square, London WC1N 3BG, or email: pals@uclh.nhs.uk

## 12. Will my information or samples be used for commercial purposes?

Successful research by us and others using your coded information and coded biological samples collected in the course of this study could result in a commercial test or therapeutic product with significant value, such as a product for the treatment of HD. You will not receive any financial benefit from such a result.





# 13. Who has reviewed this study?

All research in the NHS is looked at by an independent group of people called a Research Ethics Committee. A favourable ethical opinion has been obtained from Queen Square Research Ethics Committee. NHS Trust Management Approval has also been given.

#### 14. Insurance


The study is insured under UCL's insurance policy which provides liabilities (negligence) of UCL and its employees or agents. The policy will be renewed annually until the end of the study.

University College London holds insurance against claims from participants for harm caused by their participation in this clinical study. Participants may be able to claim compensation if they can prove that UCL has been negligent. However, if this clinical study is being carried out in a hospital, the hospital continues to have a duty of care to the participant of the clinical study. University College London does not accept liability for any breach in the hospital's duty of care, or any negligence on the part of hospital employees. This applies whether the hospital is an NHS Trust or otherwise.

#### 15. Could the study end early?

You may be withdrawn from this study if you do not follow the directions of this study or if your medical condition changes so that staying in this study might risk your health or this research. Your participation in this study may also end if the sponsor (UCL) or Principal Investigator (Prof Tabrizi) decides to terminate the study for safety or other reasons.

#### 16. How do I get in touch with the study team?

For more information concerning this research or if you believe that you have suffered a research related injury, please contact

Professor Sarah Tabrizi Box 104 National Hospital for Neurology & Neurosurgery Queen Square London WC1N 3B

Telephone 020 3108 7464, Research Team Telephone 020 3108 7483

HD Young Adult Study 2.0, EDGE (Sponsor) number: 145646, IRAS number: 303499, Control PIS/ICF, Version 2.1, 7th Sept 2023





# **HD-YAS 2.0**

(IRAS number: 303499)

| Patient identification number | |
|---|---|
| Informed consent form (CONTROL) | Please initial if you agree |
| I have read and understood the Control Information Sheet and Informed Consent Form <b>version 2.1</b> , <b>7</b> <sup>th</sup> <b>Sept 2023</b> , for the above study. I have had the opportunity to consider the information and ask questions, and have received satisfactory answers. I understand I will receive a signed copy of this informed consent document. | |
| I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | |
| I agree to undergo the 3T MRI scan and its use for research. | |
| I understand that sections of my medical notes, and data collected during the study, may be looked at by people from Prof Tabrizi's research team, sponsor, appointed service providers, regulatory authorities or the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | |
| I understand that my data will be stored with a coded research identifier to protect my identity. | |
| I understand that my coded samples and coded data will be shared with Prof Tabrizi's appointed partners from academic, not-for-profit and/or commercial research organisations and other HD researchers for research purposes. | |
| I understand that my coded samples and coded data will be shared with CHDI and by CHDI with other researchers and service providers for research purposes. | |
| I give permission for my coded data and coded samples to be shared in this way. | |
| I understand that the data generated and tissue collected during this study may be used for future commercial development of products/tests/treatments/biomarkers and I will not benefit financially from this. | |

HD Young Adult Study 2.0, EDGE (Sponsor) number: 145646, IRAS number: 303499, Control PIS/ICF, Version 2.1, 7th Sept 2023 







| I understand that data generated during the study will be sent outside of the United Kingdom where laws protecting my personal information may be different to my own country. | | |
|---|---|---|
| agree to my General Practitioner being informed of my participation in the study. | | |
| Should I lose the capacity to consent during the study, I agree to any data, DNA, blood and CSF samples (if relevant) collected prior to my withdrawal being retained and used for research related to this study and for future ethically approved research. | | |
| I give permission for the study team to contact me after HD-YAS visits to inform me of any future potential research studies or clinical trials in HD. | | |
| | Please initial box | of choice |
| Consent to optional CSF and Blood sample collection I wish to participate in the optional CSF collection part of this study and agree to provide blood samples and to undergo the lumbar puncture to collect spinal fluid. | Yes | No |
| Consent to additional MEG and 7T MRI I wish to participate in the optional MEG and 7T MRI part of this study and agree to undergo the MEG and 7T MRI scanning. | Yes No | N/A |
| I agree to take part in the above study. | Please initial if yo | ou agree |

HD Young Adult Study 2.0, EDGE (Sponsor) number: 145646, IRAS number: 303499, Control PIS/ICF, Version 2.1, 7<sup>th</sup> Sept 2023 





| Control of Destriction | D. J. J. M | D.1. |
|---|---|---|
| Signature of Participant | Printed Name | Date |
| For Study Site Staff | | |
| <b>Person Obtaining Consent.</b> I have read to form. An explanation of this study was go satisfaction. In my judgement, the partic | iven and questions were solicited and a | • |
| Signature | Printed Name D | ate |
| 1x original – into Site File; 1x copy – to Participan | t; 1x copy – into medical record | |

HD Young Adult Study 2.0, EDGE (Sponsor) number: 145646, IRAS number: 303499, Control PIS/ICF, Version 2.1, 7<sup>th</sup> Sept 2023

